CLINICAL TRIAL: NCT06770140
Title: Unraveling the Blood Microbiome in Postoperative Recurrence of Crohn's Disease
Acronym: IBDbloom
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Merel Verweij, MD, Erasmus Medical Center
Other Study IDs: 12313
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Crohn's Disease (CD)
Keywords: Ileocolonic resection; Blood microbiome; Postoperative recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, feces, biopsies and resection material
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Non-recurrence patients: Patients that do not have postoperative recurrence at colonoscopy 6 months after surgery.
- Recurrence patients: Patients that do have postoperative recurrence at colonoscopy 6 months after surgery.
- Healthy controls: Patients without Inflammatory Bowel Disease

SUMMARY:
Crohn's disease, a chronic inflammation of the gastro-intestinal tract, is a disease with a complex pathogenetic background. Hereditary factors, environmental factors and the gut flora play a varying role in its onset, however, this role remains unclear to date. We hypothesize to detect tiny fragments of microbial DNA from the gut in the bloodstream, due to disruption in the natural defences of the gut lining. If this is true, it may hold the key to understanding why Crohn's disease recurs after surgery.

Our objective in this study is to test retrospectively, if we can detect any difference in microbial DNA from the blood of ileocolonic resection (ICR) patients that do and do not show recurrence at the time of follow-up endoscopy at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's Disease
* Adult ≥ 16 years
* Undergoing an ileocolonic resection or reresection
* Written informed consent

Exclusion Criteria:

* Use of antibiotics in the past 8 weeks at the timepoints when blood is withdrawn and feces is collected.
* Use of probiotics in the past 8 weeks at the timepoints when blood is withdrawn and feces is collected.
* Not willing to collect extra biosamples

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be identified at the outpatient clinic at the dept. of gastroenterology or department of surgery or at a multidisciplinary meeting.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Differences in bloodmicrobiome between recurrence & non recurrence patients. | From enrollment to the postoperative endoscopy (at 6 months follow-up).
  To test retrospectively, if we can detect any difference in microbial DNA from the blood of ICR patients that do and do not show recurrence, defined as a Rutgeerts score ≥ i2b at the time of follow-up endoscopy at 6 months.

SECONDARY OUTCOMES:
o To identify blood biomarkers predicting postoperative recurrence in Crohn's disease. | From enrollment to the postoperative endoscopy (at 6 months follow-up).
o To identify histological parameters predicting postoperative recurrence in Crohn's disease. | From enrollment to the postoperative endoscopy (at 6 months follow-up).
o To correlate blood biomarkers with fecal biomarkers predicting postoperative recurrence in Crohn's disease. | From enrollment to the postoperative endoscopy (at 6 months follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands